CLINICAL TRIAL: NCT01921764
Title: Implementation of Physical Exercise at the Workplace (IRMA08) - Healthcare Workers
Acronym: IRMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Responsible Party: Principal Investigator, Lars L. Andersen, Professor, PhD, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRMA08
Record Dates: First submitted 2013-08-10; First posted 2013-08-13 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Workplace physical exercise (Experimental): Physical exercise (kettlebells, elastic bands, exercise balls) performed at the workplace with coaching
  Interventions: Behavioral: Workplace physical exercise
- Home physical exercise (Active Comparator): Physical exercise performed at home with elastic bands and bodyweight exercises with instruction to follow the exercises at http://www.jobogkrop.dk/Oevelser-til-nakke-og-ryg/Oevelser
  Interventions: Behavioral: Home physical exercise

INTERVENTIONS:
Behavioral: Workplace physical exercise
  Arms: Workplace physical exercise
Behavioral: Home physical exercise
  Arms: Home physical exercise

SUMMARY:
The prevalence and consequences of musculoskeletal pain is considerable among healthcare workers, allegedly due to high physical work demands of healthcare work. Previous studies have shown promising results of physical exercise for relieving pain among different occupational groups, but the question remains whether such physical exercise should be performed at the workplace or in the private sphere at home. Performing physical exercise at the workplace together with colleagues may be more motivating for some employees and thus increase compliance. On the other hand, physical exercise at the workplace may be costly for the employers in terms of time spend. Thus, relevant ground exists to compare the efficacy of workplace- versus home-based training on musculoskeletal pain. This study investigates the effect of workplace-based versus home-based physical exercise on musculoskeletal pain among healthcare workers.

The main hypothesis is that physical exercise at the workplace for 10 weeks compared with physical exercise at home results in reduced musculoskeletal pain among healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* healthcare worker
* female
* age 18-67

Exclusion Criteria:

* life threatening disease
* pregnancy

Ages: 18 Years to 67 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | change from baseline to week 10
  The change in "pain intensity during the last week" from baseline to 10 week follow-up between the workplace- and home-training group. The home-training group will be considered the reference group. 2-way analysis of variance (Proc Mixed of SAS) with repeated measures will be used, with time and group as fixed factors and subject as random factor. Department will be added as a cluster effect.

SECONDARY OUTCOMES:
Muscle function | change from baseline to week 10
Work ability index (WAI) | change from baseline to week 10
Physical exertion during work | change from baseline to week 10

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

REFERENCES:
- [Derived] Jakobsen MD, Sundstrup E, Brandt M, Andersen LL. Psychosocial benefits of workplace physical exercise: cluster randomized controlled trial. BMC Public Health. 2017 Oct 10;17(1):798. doi: 10.1186/s12889-017-4728-3. PMID 29017479
- [Derived] Jakobsen MD, Sundstrup E, Brandt M, Jay K, Aagaard P, Andersen LL. Physical exercise at the workplace prevents deterioration of work ability among healthcare workers: cluster randomized controlled trial. BMC Public Health. 2015 Nov 25;15:1174. doi: 10.1186/s12889-015-2448-0. PMID 26607232
- [Derived] Jakobsen MD, Sundstrup E, Brandt M, Jay K, Aagaard P, Andersen LL. Effect of Workplace- versus Home-Based Physical Exercise on Muscle Response to Sudden Trunk Perturbation among Healthcare Workers: A Cluster Randomized Controlled Trial. Biomed Res Int. 2015;2015:902896. doi: 10.1155/2015/902896. Epub 2015 Oct 25. PMID 26583145
- [Derived] Jakobsen MD, Sundstrup E, Brandt M, Kristensen AZ, Jay K, Stelter R, Lavendt E, Aagaard P, Andersen LL. Effect of workplace- versus home-based physical exercise on pain in healthcare workers: study protocol for a single blinded cluster randomized controlled trial. BMC Musculoskelet Disord. 2014 Apr 7;15:119. doi: 10.1186/1471-2474-15-119. PMID 24708570